CLINICAL TRIAL: NCT03232203
Title: Evaluation of Referring HCPs' and Parents'/Carers' Understanding of Specific Risks Associated With Strimvelis™ Treatment
Brief Title: Evaluating the Effectiveness of STRIMVELIS Risk Minimization Measures (RMMs)
Status: Completed | Type: Observational
Sponsor: Fondazione Telethon (Other)
Responsible Party: Sponsor
Other Study IDs: STRIM-001
Record Dates: First submitted 2017-07-25; First posted 2017-07-27 (Actual); Last update posted 2023-11-14 (Actual); Status verified 2023-11

CONDITIONS: Severe Combined Immunodeficiency Due to ADA Deficiency
Keywords: Human leukocyte antigen; Key Risk Message; ADA-SCID; Health care providers
MeSH Terms: conditions — Severe combined immunodeficiency due to adenosine deaminase deficiency

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Health care providers: A HCP survey instrument of approximately 20 questions will be provided. Survey questions will be based on the STRIMVELIS summary of product characteristics and educational materials
  Interventions: Drug: STRIMVELIS
- Parent/carer: A parent/carer survey instrument of approximately 20 questions will be provided. Survey questions will be based on the STRIMVELIS Patient Information Leaflet and educational materials
  Interventions: Drug: STRIMVELIS

INTERVENTIONS:
Drug: STRIMVELIS — It is the Autologous cluster of differentiation (CD) 34+ enriched cell fraction that contains CD34+ cells transduced with retroviral vector that encodes for the human ADA complementary Deoxyribonucleic acid (cDNA) sequence. HCP who have previously referred a patient for STRIMVELIS treatment or a parent's/carer's child who previously received treatment with STRIMVELIS will be recruited to the study

SUMMARY:
STRIMVELIS is a medicinal product that restores adenosine deaminase (ADA) function in hematopoietic cell lineages, thereby preventing impaired immune function. STRIMVELIS is indicated for the treatment of patients with ADA- severe combined immunodeficiency (SCID), for whom suitable human leukocyte antigen (HLA)-matched related stem cell donor is not available. The objective of this study is to evaluate the effectiveness of routine and additional risk minimization measures by assessing the understanding of referring health care providers (HCPs) and parents/carers (hereby referred as participants) with regard to the specific risks associated with STRIMVELIS. In this cross-sectional study, surveys will be provided to referring HCPs and parents/carers of children approximately six months after treatment with STRIMVELIS. The study will recruit for approximately two years or until a maximum of 10 referring HCPs and 10 parents/carers have completed their respective surveys, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* HCPs or HCPs' close family members may not have been employees of Orchard, Pharmaceutical Product Development, LLC (PPD), the Food and Drug Administration (FDA), or the European Medicines Agency (EMA).
* HCPs must be licensed
* An HCP must not have previously completed a survey regarding STRIMVELIS educational materials.
* An HCP must have previously referred a patient for STRIMVELIS treatment.
* Parents/carers or parents'/carers' close family members may not have been employees of Orchard, PPD, FDA, or EMA.
* A parent/carer must not have previously completed a survey regarding STRIMVELIS educational materials.
* A parent's or carer's child must have previously received treatment with STRIMVELIS

Exclusion Criteria:

* No exclusion criteria

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Parents/carers and referring HCPs of patients enrolled within this registry or patients treated with STRIMVELIS outside of the registry will be contacted separately and asked to participate in their respective surveys evaluating the effectiveness of risk minimization measures.
Sampling Method: Probability Sample
Enrollment: 16 (Actual)
Dates: Start 2018-04-12 (Actual); Primary Completion 2021-06-25 (Actual); Study Completion 2021-06-25 (Actual)

PRIMARY OUTCOMES:
Proportion of HCPs providing the correct response | Up to 2 years
  A series of questions concerning the specific risks associated with STRIMVELIS will be asked during survey. Data from all survey respondents will be analyzed and reported as descriptive statistics.
Proportion of Parents/Carers providing the correct response | Up to 2 years
  A series of questions concerning the specific risks associated with STRIMVELIS will be asked during survey. Data from all survey respondents will be analyzed and reported as descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Fondazione Telethon, Study Director — Fondazione Telethon
Locations (1):
- Ospedale San Raffaele - Telethon Institute for Gene Therapy (OSR-TIGET), Milan, Italy